CLINICAL TRIAL: NCT00117338
Title: A Multicenter, Randomized, Double-Blind Study Comparing the Clinical Effects of Intravenous Montelukast With Placebo in Pediatric Patients (Ages 6 to 14 Years) With Acute Asthma
Brief Title: A Study of an Intravenous Drug in Pediatric Patients With Acute Asthma (0476-301)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0476-301; MK0476-301; 2005_026
Record Dates: First submitted 2005-06-30; First posted 2005-07-06 (Estimated); Results first posted 2009-08-11 (Estimated); Last update posted 2024-05-10 (Actual); Status verified 2022-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: placebo (unspecified)
- 2 (Active Comparator): montelukast sodium
  Interventions: Drug: montelukast sodium

INTERVENTIONS:
Drug: montelukast sodium — Montelukast IV 5.25 mg lyophilized (reconstituted in 20 mL of 3.3% dextrose/0.3% sodium chloride) for a study approximately 120 minutes in duration
  Other Names: MK0476; SINGULAIR®
  Arms: 2
Drug: Comparator: placebo (unspecified) — Pbo for a study approximately 120 minutes in duration
  Arms: 1

SUMMARY:
This study will attempt to find out if the addition of an intravenous form of a drug that is already used for treating asthma in children will help resolve asthma attacks faster than using the current standard care alone.

DETAILED DESCRIPTION:
The duration of treatment is a one time dose.

ELIGIBILITY:
Inclusion Criteria:

* Children 6-14 years of age seeking treatment in emergency departments with acute asthma attacks

Exclusion Criteria:

* Other respiratory conditions (including congenital lung abnormalities) or other acute illnesses that would complicate current treatment and response for asthma

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 276 (Actual)
Dates: Start 2005-07; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morris CR, Becker AB, Pinieiro A, Massaad R, Green SA, Smugar SS, Gurner DM. A randomized, placebo-controlled study of intravenous montelukast in children with acute asthma. Ann Allergy Asthma Immunol. 2010 Feb;104(2):161-71. doi: 10.1016/j.anai.2009.11.065. PMID 20306820

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase III World Wide (U.S., Europe, Asia, South America, and Lithuania) Multicenter Study. Study Start Date: July 2005 Primary Completion Date: March 2008 Study Completion Date: March 2008
Period: Overall Study
Arm/Group | Montelukast Intravenous (IV) 5.25 mg | Placebo
Started | 145 | 131
Completed | 140 | 127
Not Completed | 5 | 4
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 3 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Did not meet Inclusion Criteria | 1 | 0
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Montelukast Intravenous (IV) 5.25 mg | Placebo | Total
Number analyzed (Participants) | 145 | 131 | 276
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.2 (2.36) | 8.9 (2.32) | 9.1 (2.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 50 | 105
  Male | 90 | 81 | 171
Race/Ethnicity [Number; unit: participants]
  White (Non-Hispanic) | 16 | 16 | 32
  Black | 18 | 16 | 34
  Hispanic | 59 | 53 | 112
  Asian | 18 | 18 | 36
  Multi-Racial | 34 | 27 | 61
  Other | 0 | 1 | 1
Baseline FEV 1 (L) [Mean (Standard Deviation); unit: Liters] — Forced Expiratory Volume in one second, measured in Liters (FEV 1 (L))
  A total of 4/276 (1-montelukast; 3-placebo) randomized patients were excluded from the Full Analysis Set (FAS) of the primary endpoint
  Liters | 1.06 (0.5) | 1.00 (0.5) | 1.0 (0.5)
Baseline FEV1 (Percent predicted) [Mean (Standard Deviation); unit: Percent] — Percent of predicted baseline Forced Expiratory Volume in one second (FEV1)
  A total of 4/276 (1-montelukast; 3-placebo) randomized patients were excluded from the Full Analysis Set (FAS) of the primary endpoint
  Percent | 51.8 (16.8) | 50.6 (17.4) | 51.2 (17.1)

OUTCOME MEASURES:

1. Primary Outcome: Improvement in FEV1 (Forced Expiratory Volume in 1 Second) Over the First 60 Minutes After Administration
Description: Improvement in FEV1 as the time-weighted average change from baseline over 60 minutes following the end of study drug administration. Time-weighted average of the changes from baseline obtained over the 60 minutes (at 60, 45, 30 and 15) with the time interval between any measurement and the measurement prior to it used as the weighting factor.
Time Frame: Baseline and (time weighted average over) 60 Minutes
Population: Full Analysis Set (FAS). The FAS population includes all randomized patients who received double-blind study drug, and with efficacy measurements both at baseline and at least one time point over the time interval considered.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Montelukast Intravenous (IV) 5.25 mg | Placebo
Number analyzed (Participants) | 144 | 128
Liters | 0.08 [0.02 to 0.13] | 0.07 [0.01 to 1.12]
Statistical Analysis 1: Comparison: Montelukast Intravenous (IV) 5.25 mg vs Placebo; Test type: Superiority or Other; p = 0.775, ANCOVA; Model terms: treatment, region (US, non-US) and baseline FEV1 as covariate; Mean Difference (Final Values) = 0.01, 95% CI [-0.06 to 0.08]

2. Secondary Outcome: Change From Baseline in Modified Pulmonary Index [mPI] Score
Description: Change from baseline in modified pulmonary index [mPI] score assessed 60 minutes following the end of study drug administration. mPI questionnaire scores each component on a scale of 0 to 3 (low to high) with a total possible score of 12.
  The components are respiratory rate, wheezing, prolongation of expiration (Inspiratory:Expiratory ratio), and accessory muscle use.
Time Frame: Baseline and 60 minutes
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Montelukast Intravenous (IV) 5.25 mg | Placebo
Number analyzed (Participants) | 143 | 128
Score on a scale | -2.95 [-3.26 to -2.63] | -2.96 [-3.29 to -2.63]
Statistical Analysis 1: Comparison: Montelukast Intravenous (IV) 5.25 mg vs Placebo; Test type: Superiority or Other; p = 0.931, ANCOVA; Model terms: treatment, region (US, non-US) and baseline FEV1 as covariate; Mean Difference (Final Values) = 0.02, 95% CI [-0.41 to 0.45]

3. Secondary Outcome: Number of Participants With Treatment Failure (Hospitalization or Time to Decision to Discharge > 2 Hours)
Description: Treatment Failure is defined as a.) patients who required hospitalization, or b.) patients for whom a decision to discharge home has not been reached by 2 hours following the end of study drug administration.
Time Frame: 120 minutes
Population: Full Analysis Set (FAS). At least one post-randomization measurement obtained subsequent to at least one dose of study treatment was required for inclusion in the analysis of treatment failure endpoint. Baseline FEV1 measurement was also required to assess this endpoint since it was included in the model.
Measure: Number; unit: Participants
Arm/Group | Montelukast Intravenous (IV) 5.25 mg | Placebo
Number analyzed (Participants) | 144 | 128
Participants
  Hospitalization | 28 | 33
  Decision to Discharge Home not Reached by 2 Hours | 37 | 26
Statistical Analysis 1: Comparison: Montelukast Intravenous (IV) 5.25 mg vs Placebo; Test type: Superiority or Other; p = 0.975, Regression, Logistic; Model terms: treatment and baseline FEV1 as covariate; Odds Ratio (OR) = 0.99, 95% CI [0.61 to 1.61]

4. Secondary Outcome: Time-Weighted Average Change in FEV1 Over 45 Minutes Following the End of Study Drug Administration
Description: Improvement in FEV1 as time-weighted average change from baseline over 45 minutes following the end of study drug administration: Time-weighted average of the changes from baseline obtained over the 45 minutes (at 45, 30 and 15) with the time interval between any measurement and the measurement prior to it used as the weighting factor.
Time Frame: Baseline and (time-weighed average over) 45 Minutes
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Montelukast Intravenous (IV) 5.25 mg | Placebo
Number analyzed (Participants) | 142 | 127
Liters | 0.07 [0.02 to 0.12] | 0.05 [0.00 to 0.11]
Statistical Analysis 1: Comparison: Montelukast Intravenous (IV) 5.25 mg vs Placebo; Test type: Superiority or Other; p = 0.612, ANCOVA; Model terms: treatment, region (US, non-US) and baseline FEV1 as covariate; Mean Difference (Final Values) = 0.02, 95% CI [-0.05 to 0.09]

5. Secondary Outcome: Time-Weighted Average Change in FEV1 Over 30 Minutes Following the End of Study Drug Administration
Description: Improvement in FEV1 as the time-weighted average change from baseline over 30 minutes following the end of study drug administration. Time-weighted average of the changes from baseline obtained over the 30 minutes (at 30 and 15) with the time interval between any measurement and the measurement prior to it used as the weighting factor.
Time Frame: Baseline and (time-weighted average over) 30 Minutes
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Montelukast Intravenous (IV) 5.25 mg | Placebo
Number analyzed (Participants) | 140 | 125
Liters | 0.06 [0.01 to 0.12] | 0.05 [-0.00 to 0.11]
Statistical Analysis 1: Comparison: Montelukast Intravenous (IV) 5.25 mg vs Placebo; Test type: Superiority or Other; p = 0.774, ANCOVA; Model terms: treatment, region (US, non-US) and baseline FEV1 as covariate; Mean Difference (Final Values) = 0.01, 95% CI [-0.06 to 0.08]

6. Secondary Outcome: Change in FEV1 After 15 Minutes Following the End of Study Drug Administration
Description: Improvement in FEV1 as the time-weighted average change from baseline over the first 15 minutes following the end of study drug administration. Change = 15 minutes value minus Baseline value
Time Frame: Baseline and 15 Minutes
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Montelukast Intravenous (IV) 5.25 mg | Placebo
Number analyzed (Participants) | 121 | 115
Liters | 0.06 [0.01 to 0.10] | 0.01 [-0.03 to 0.06]
Statistical Analysis 1: Comparison: Montelukast Intravenous (IV) 5.25 mg vs Placebo; Test type: Superiority or Other; p = 0.173, ANCOVA; Model terms: treatment, region (US, non-US) and baseline FEV1 as covariate; Mean Difference (Final Values) = 0.04, 95% CI [-0.02 to 0.11]

7. Secondary Outcome: Total Dose of β-agonist Administered Per Patient Over a Period of 2 Hours Following the End of Study Drug Administration
Description: Median total dose of β-agonist administered per patient over a period of 2 hours following the end of study drug administration.
Time Frame: 120 minutes
Population: At least one post-randomization measurement obtained subsequent to at least one dose of study treatment was required for inclusion in the analysis of total doses of Beta-Agonist (mg) endpoint.
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Montelukast Intravenous (IV) 5.25 mg | Placebo
Number analyzed (Participants) | 144 | 127
mg | 1.0 [0.0 to 4.3] | 0.6 [0.0 to 3.8]
Statistical Analysis 1: Comparison: Montelukast Intravenous (IV) 5.25 mg vs Placebo; Test type: Superiority or Other; p = 0.580, ANCOVA; ANCOVA model (Nonparametric) based on Tukey's normalized ranks with terms treatment, region (US, non-US) and baseline FEV1 as covariate

ADVERSE EVENTS:
Arm/Group | Montelukast Intravenous (IV) 5.25 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 2 | 2
Other Adverse Events (participants affected / at risk) | 20 | 21
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Montelukast Intravenous (IV) 5.25 mg | Placebo
Any Infections And Infestations (Infections and infestations) | 1/145 | 0/131
Pneumonia (Infections and infestations) | 1/145 | 0/131
Any Injury, Poisoning And Procedural Complications (Injury, poisoning and procedural complications) | 0/145 | 1/131
Overdose (Injury, poisoning and procedural complications) | 0/145 | 1/131
Any Respiratory, Thoracic And Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 2/145 | 1/131
Asthma (Respiratory, thoracic and mediastinal disorders) | 0/145 | 1/131
Asthmatic Crisis (Respiratory, thoracic and mediastinal disorders) | 2/145 | 0/131
OTHER ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Montelukast Intravenous (IV) 5.25 mg | Placebo
Any Cardiac Disorders (Cardiac disorders) | 1/145 | 0/131
Tachycardia (Cardiac disorders) | 1/145 | 0/131
Any Gastrointestinal Disorders (Gastrointestinal disorders) | 5/145 | 6/131
Abdominal Pain (Gastrointestinal disorders) | 0/145 | 1/131
Abdominal Pain Upper (Gastrointestinal disorders) | 2/145 | 0/131
Constipation (Gastrointestinal disorders) | 0/145 | 1/131
Diarrhoea (Gastrointestinal disorders) | 1/145 | 1/131
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1/145 | 0/131
Nausea (Gastrointestinal disorders) | 1/145 | 1/131
Vomiting (Gastrointestinal disorders) | 1/145 | 2/131
Any General Disorders And Administration Site Conditions (General disorders) | 2/145 | 1/131
Chest Pain (General disorders) | 1/145 | 0/131
Infusion Site Extravasation (General disorders) | 0/145 | 1/131
Infusion Site Pain (General disorders) | 1/145 | 0/131
Any Infections And Infestations (Infections and infestations) | 5/145 | 5/131
Bronchitis Bacterial (Infections and infestations) | 1/145 | 0/131
Gastroenteritis (Infections and infestations) | 1/145 | 0/131
Influenza (Infections and infestations) | 0/145 | 1/131
Nasopharyngitis (Infections and infestations) | 1/145 | 2/131
Pharyngitis (Infections and infestations) | 1/145 | 0/131
Rhinitis (Infections and infestations) | 0/145 | 1/131
Sinusitis (Infections and infestations) | 0/145 | 2/131
Tonsillitis (Infections and infestations) | 1/145 | 0/131
Any Musculoskeletal And Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 1/145 | 1/131
Arthralgia (Musculoskeletal and connective tissue disorders) | 0/145 | 1/131
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1/145 | 0/131
Any Nervous System Disorders (Nervous system disorders) | 6/145 | 2/131
Dizziness (Nervous system disorders) | 0/145 | 1/131
Headache (Nervous system disorders) | 5/145 | 1/131
Syncope Vasovagal (Nervous system disorders) | 1/145 | 0/131
Any Respiratory, Thoracic And Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 5/145 | 9/131
Asthma (Respiratory, thoracic and mediastinal disorders) | 4/145 | 7/131
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1/145 | 0/131
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0/145 | 2/131
Any Skin And Subcutaneous Tissue Disorders (Skin and subcutaneous tissue disorders) | 0/145 | 2/131
Prurigo (Skin and subcutaneous tissue disorders) | 0/145 | 1/131
Pruritus (Skin and subcutaneous tissue disorders) | 0/145 | 1/131
Any Vascular Disorders (Vascular disorders) | 0/145 | 1/131
Diastolic Hypotension (Vascular disorders) | 0/145 | 1/131

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.